CLINICAL TRIAL: NCT06145906
Title: Application Value of Whole-procedure Optimization for Catheter Ablation of Atrial Fibrillation
Status: Recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HenanPPH Cardiology
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; optimized strategies and workflows
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paroxysmal AF group: AF that terminates spontaneously or with intervention within 7 days of onset
  Interventions: Procedure: Pulmonary vein isolation plus superior vena cava isolation
- Persistent AF group: AF that is continuously sustained beyond 7 days, including episodes terminated by cardioversion (drugs or electrical cardioversion) after ≥7 days
  Interventions: Procedure: PVI, superior vena cava isolation, and linear ablation of linear ablations of the mitral isthmus, roofline and posterior wall line of the left atrium, and cavotricuspid isthmus

INTERVENTIONS:
Procedure: Pulmonary vein isolation plus superior vena cava isolation — Pulmonary vein isolation plus superior vena cava isolation
  Groups: Paroxysmal AF group
Procedure: PVI, superior vena cava isolation, and linear ablation of linear ablations of the mitral isthmus, roofline and posterior wall line of the left atrium, and cavotricuspid isthmus — PVI, superior vena cava isolation, and linear ablation of linear ablations of the mitral isthmus, roofline and posterior wall line of the left atrium, and cavotricuspid isthmus
  Groups: Persistent AF group

SUMMARY:
The success rate of single-procedure atrial arrhythmia-free survival particularly ranged from 40% to 66% in persistent AF ablation. However, The surgical Cox maze III procedure has been established to be an effective curative strategy for AF with an AF-free survival rate of more than 95%. The main reason is the difficulty of creating continuous, transmural, and durable lesions by catheter ablation, especially when the procedure is performed on some complex anatomical structures in which epicardial muscular bundles may serve as components of the reentrant circuits.

The durability of the conduction block is a crucial factor for long-term effective AF ablation since previous studies reported that the reconnected Pulmonary veins contributed to the atrial tachycardia recurrence after persistent AF ablation. In addition, it is possible that the inadequate lesions accidentally produce new arrhythmogenic substrates. Therefore, new and better techniques are always chosen to minimize the reconnection of Pulmonary vein isolation (PVI) and additional ablation.

For paroxysmal AF, the ablation strategy of PVI plus superior vena cava isolation is chosen while PVI, superior vena cava isolation, and linear ablation of linear ablations of the mitral isthmus, roofline and posterior wall line of the left atrium, and cavotricuspid isthmus (CTI) for persistent AF. Any symptomatic or asymptomatic atrial arrhythmia lasting more than 30 seconds was regarded as an AF recurrence after a 3-month blanking period. The primary outcome was defined as 12-month atrial arrhythmia-free survival. The secondary outcomes include the block rate of PVI, superior vena cava isolation, and all linear ablations.

ELIGIBILITY:
Inclusion Criteria:

* Radiofrequency catheter ablation for the first time
* AF rhythm recorded by ECG

Exclusion Criteria:

* Thrombosis in left atrium
* Left ventricular ejection fraction of < 35%
* Abnormal thyroid function
* Previous history of AF radiofrequency ablation and CABG
* Left atrium diameter of > 65 mm or the volume of > 200 ml

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are ECG which can be definitely diagnosed as atrial fibrillation, that is: P wave disappeared, replaced by F wave, frequency 350-600 times / min, QRS wave rhythm is absolutely irregular, RR interval is uneven, QRS wave shape is normal
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
AF recurrence | 12 months
  Any symptomatic or asymptomatic atrial arrhythmia lasting more than 30 seconds after a 3-month blanking period

SECONDARY OUTCOMES:
initial block rate | intraoperation
  initial block rate of pulmonary veins isolation, superior vena cava isolation and additional ablation lines

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL. Corrigendum to: 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Oct 21;42(40):4194. doi: 10.1093/eurheartj/ehab648. No abstract available. PMID 34520521
- [Background] El Haddad M, Taghji P, Phlips T, Wolf M, Demolder A, Choudhury R, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Determinants of Acute and Late Pulmonary Vein Reconnection in Contact Force-Guided Pulmonary Vein Isolation: Identifying the Weakest Link in the Ablation Chain. Circ Arrhythm Electrophysiol. 2017 Apr;10(4):e004867. doi: 10.1161/CIRCEP.116.004867. PMID 28381417
- [Result] Mark DB, Anstrom KJ, Sheng S, Piccini JP, Baloch KN, Monahan KH, Daniels MR, Bahnson TD, Poole JE, Rosenberg Y, Lee KL, Packer DL; CABANA Investigators. Effect of Catheter Ablation vs Medical Therapy on Quality of Life Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1275-1285. doi: 10.1001/jama.2019.0692. PMID 30874716
- [Result] Mont L, Bisbal F, Hernandez-Madrid A, Perez-Castellano N, Vinolas X, Arenal A, Arribas F, Fernandez-Lozano I, Bodegas A, Cobos A, Matia R, Perez-Villacastin J, Guerra JM, Avila P, Lopez-Gil M, Castro V, Arana JI, Brugada J; SARA investigators. Catheter ablation vs. antiarrhythmic drug treatment of persistent atrial fibrillation: a multicentre, randomized, controlled trial (SARA study). Eur Heart J. 2014 Feb;35(8):501-7. doi: 10.1093/eurheartj/eht457. Epub 2013 Oct 17. PMID 24135832
- [Result] Inoue K, Hikoso S, Masuda M, Furukawa Y, Hirata A, Egami Y, Watanabe T, Minamiguchi H, Miyoshi M, Tanaka N, Oka T, Okada M, Kanda T, Matsuda Y, Kawasaki M, Hayashi K, Kitamura T, Dohi T, Sunaga A, Mizuno H, Nakatani D, Sakata Y; OCVC Arrhythmia Investigators. Pulmonary vein isolation alone vs. more extensive ablation with defragmentation and linear ablation of persistent atrial fibrillation: the EARNEST-PVI trial. Europace. 2021 Apr 6;23(4):565-574. doi: 10.1093/europace/euaa293. PMID 33200213
- [Result] Yu HT, Shim J, Park J, Kim IS, Kim TH, Uhm JS, Joung B, Lee MH, Kim YH, Pak HN. Pulmonary Vein Isolation Alone Versus Additional Linear Ablation in Patients With Persistent Atrial Fibrillation Converted to Paroxysmal Type With Antiarrhythmic Drug Therapy: A Multicenter, Prospective, Randomized Study. Circ Arrhythm Electrophysiol. 2017 Jun;10(6):e004915. doi: 10.1161/CIRCEP.116.004915. PMID 28611206
- [Result] Shah S, Barakat AF, Saliba WI, Abdur Rehman K, Tarakji KG, Rickard J, Bassiouny M, Baranowski B, Tchou P, Bhargava M, Chung M, Dresing T, Callahan T, Cantillon D, Kanj M, Lindsay BD, Wazni OM, Hussein AA. Recurrent Atrial Fibrillation After Initial Long-Term Ablation Success: Electrophysiological Findings and Outcomes of Repeat Ablation Procedures. Circ Arrhythm Electrophysiol. 2018 Apr;11(4):e005785. doi: 10.1161/CIRCEP.117.005785. PMID 29654129